CLINICAL TRIAL: NCT05559398
Title: Glenzocimab for REperfusion in the Setting of Endovascular Therapy for Brain infarctioN: GREEN Study
Acronym: GREEN
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP 201028 / ACT-CS-004; 2021-000889-16 (EudraCT Number)
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Stroke, Acute; Stroke, Ischemic
Keywords: Platelet glycoprotein VI; Endovascular therapy
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — glenzocimab

STUDY DESIGN:
Intervention Model Description: Randomized, double blinded, multicentre, placebo controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Glenzocimab (Experimental)
  Interventions: Drug: Glenzocimab

INTERVENTIONS:
Drug: Glenzocimab — Glenzocimab (ACT-017, Acticor Biotech) is formulated for IV administration as a sterile product with 20 mM sodium citrate and 130 mM sodium chloride buffer at pH of 5.0.
  It is supplied for clinical trial use in vials containing 50 mL of the drug product at a concentration of 10 mg/mL.
  Each vial contains 500 mg of glenzocimab. Two vials (2x500 mg) of glenzocimab should be administered concomitantly for eligible patients for a total daily dose of 1g.
  Glenzocimab is intended to be administered as an IV infusion over 6 hrs, with 1/4 of the dose administered by a 15-minute bolus and 3/4 of the dose administered by 5h45min-slow infusion.
  Arms: Glenzocimab
Drug: Placebo — Placebo of glenzocimab is 0.9%NaCl (Acticor Biotech) for IV administration. It is supplied for clinical trial use in vials of 50 mL. Two vials of placebo of glenzocimab should be administered concomitantly for eligible patients.
  Arms: Placebo

SUMMARY:
Emergent reperfusion is the main goal for acute ischemic stroke therapy (AIS). Endovascular therapy (EVT) is recommended within 6 hrs of stroke onset, and up to 24 hrs following perfusion imaging criteria.

Despite the major benefit associated with MT, more than 50% of the patients remain disabled at 3 months. Reperfusion rates after MT are critical to determine functional outcome. However, complete reperfusion is obtained in only 50 % of the patients, due to, at least in part, erratic emboli and/or no-reflow processes. The aim of this study is to evaluate the efficacy of glenzocimab in addition to EVT and compared to EVT plus placebo, whether or not associated with ntravenous thrombolysis (IVT), on functional outcome at day 90.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older (Age≥18 years)
2. No significant pre-stroke disability (pre-stroke mRS must be equal to 0 or 1);
3. Indication of EVT within the time-window of 0 to 24 hrs in participants treated with or without intravenous thrombolysis;
4. Participants presenting with a target mismatch defined by an initial infarct volume (ischemic core) of less than 70 ml, a ratio of volume of ischemic tissue to initial infarct volume of 1.8 or more, and an absolute volume of potentially reversible ischemia (penumbra) of 15 ml or more on magnetic resonance imaging (MRI) or, when this is not possible, on perfusion computed tomography (CTP);
5. Occlusion of the cervical or intracranial internal carotid artery (ICA) or the proximal middle cerebral artery (MCA - M1 and M2), on magnetic resonance angiography (MRA) or, when this is not possible, on CT angiography (CTA);
6. Informed consent signed:

   * By the patient
   * Or informed consent signed by a family members/trustworthy person if his condition does not allow him to express his consent by written as per L. 1111-6,
   * In a situation urgently and in the absence of family members/trustworthy person, the patient can be enrolled. The consent to participate to the research will be requested as soon as the condition of the patient will allow him to consent.
7. Post-menopausal women defined as not having menses for 12 months without an alternative medical cause. For WOCBP, a highly effective birth control method should be in place that can achieve a failure rate of less than 1% per year that should last for at least 2 months after IMP administration.

   Birth control methods which may be considered as highly effective in WOCBP include:
   * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (intravaginal, transdermal),
   * progestogen-only hormonal contraception associated with inhibition of ovulation (injectable, implantable)
   * intrauterine device (IUD),
   * intrauterine hormone-releasing system (IUS),
   * bilateral tubal occlusion,
   * vasectomized partner,

   Birth control methods which may be considered as highly effective for men and that should last for 4 months after IMP administration include:
   * vasectomy,
   * use of condom combined with a highly effective birth control method for their WOCB partner.

   Please note that hormonal contraception is a risk factor for thromboembolic events and attention should be called to reconsider it passed the acute stroke phase.
8. Women of child-bearing potential must have negative results of a plasma pregnancy test (serum betaHCG).
9. Affiliation to social security or any health insurance

Exclusion Criteria:

1. Contraindications to EVT;
2. Contraindication to contrast agents
3. Pre-existing neurologic and psychiatric disease with mRS ≥ 3;
4. Unknown symptom's onset;
5. Patients under or needing immediate DAPT administration;
6. Patients previously treated by tenecteplase within 24 hrs;
7. Significant mass effect with midline shift as confirmed on CT/MRI;
8. Gastrointestinal or urinary tract hemorrhage in previous 21 days;
9. Patient with intracranial haemorrhage
10. Platelet count <100 000 mm3;
11. Pregnant or breastfeeding woman;
12. Known hypersensitivity to glenzocimab or to any of the excipients;
13. Severe renal insufficiency (Grades 4-5) with a glomerular filtration rate < 30mL/Min/1.73m2;
14. Participation in another interventional clinical trial within 30 days prior to the inclusion.
15. Persons deprived of their liberty by a judicial or administrative decision, persons subject to psychiatric care under sections L.3212-1 et L.3213-1 and persons admitted to a health or social institution for purposes other than research (L.1121-6)
16. Adults subject to a legal protection measure (L.1121-8)
17. The patient or his/her family (if the patient is unable to give his/her opinion) expresses an inability to return for protocol visits
18. patients receiving anticoagulants, as already mentioned in the non-authorized concomitant treatments
19. patients who have already received another humanized fragment of monoclonal antibody with a suspicion of hypersensitivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2022-10-10 (Estimated); Primary Completion 2025-10-10 (Estimated); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
Efficacy mRS 90 | 90 days
  The primary efficacy endpoint is the functional outcome assessed by the modified Rankin Scale (mRS) at day 90 +/- 15 days.
  The Modified Rankin Scale (mRS) is used to measure the degree of disability in patients who have had a stroke. The scale runs from 0-6, running from perfect health without symptoms to death.
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.

SECONDARY OUTCOMES:
Favorable functional outcome | 90 days
  Favorable functional outcome defined by a mRS ≤ 2 at day 90 +/- 15 days
Severe handicap | 90 days
  Proportion of patients with a severe handicap: mRS equal to 4, 5 or 6 at day 90 +/- 15 days
Survival | 90 days and 1 year
  Overall survival at 90 days and 1 year
Early reperfusion outcomes : volume | 24 hours
  Stroke volume by MRI at 24 hrs
Early reperfusion outcomes : eTICI | 24 hours
  Reperfusion at the end of procedure assessed by the expanded treatment in cerebral infarction (eTICI) score.The eTICI is defined as follows :
  grade 0: no perfusion noted (0% reperfusion) grade 1: reduction in thrombus but without any resultant filling of distal arterial branches grade 2a: reperfusion of 1-49% of the territory grade 2b50: reperfusion of 50-66% of the territory grade 2b67: reperfusion of 67-89% of the territory grade 2c: extensive reperfusion of 90-99% of the territory grade 3: complete or full reperfusion (100% reperfusion)
Early reperfusion outcomes NIHSS | 24 hours
  Early neurological improvement by National Institutes of Health Stroke Scale, or NIH Stroke Scale (NIHSS) at 24 hrs.
  The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
Quality of life | 90 days and 1 year
  EQ5D-5L at day 90 and at 1 year. EQ-5D is a standardised measure of health-related quality of life. The EQ-5D-5L descriptive system uses five dimensions. The five levels in each dimension are worded as (1) 'not /no problems', (2) 'slight problems', (3) 'moderate problems', (4) 'severe problems', and (5) 'unable to' (mobility, self-care, usual activities), 'extreme' (pain/depression), or 'extremely' (anxiety/depression). EQ-5D-5L is the sum of the five dimensions.
IntraCranial Hemorrhages | 24 hours
  Incidence of symptomatic or non-symptomatic IntraCranial Hemorrhages (ICH) at 24 hrs
Symptomatic IntraCranial Hemorrhages | 24 hours
  Incidence of symptomatic IntraCranial Hemorrhages (ICH) at 24 hrs
Non-Symptomatic IntraCranial Hemorrhages | 24 hours
  Incidence of non-symptomatic IntraCranial Hemorrhages (ICH) at 24 hrs
Adverse event | 24 hours, 7 days, 30 days, 90 days
  Incidence, nature and severity of Adverse Events, SAEs, SUSARs, Bleeding-Related Events (BREs) and/or Treatment-Emergent Adverse Events (TEAEs), at 24 hrs, at D7/discharge, 30 days and 90 days
Bleeding relating events | 90 days
  Incidence of bleeding-related events at 90 days
Anti-glenzocimab antibodies | 3 months
  Anti-glenzocimab antibodies (ADA) blood concentration at 3 months for 50 patients.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mazighi M, Lambert J, Gory B, Seners P, Calviere L, Cho TH, Aghetti A, Pasi M, Boulouis G, Lapergue B, Consoli A, Turc G, Rouchaud A, Wolff V, Pop R, Suissa L, Richard S, Cordonnier C, Arquizan C, Costalat V, Guedon A, Cognard C, Mameri L, Escalard S, Redjem H, Smajda S, Robichon E, Al Raaisi A, Boisseau W, Blanc R, Maier B, Boursin P, Dubus E, Desilles JP, Piotin M, Rigon MR, Olivot JM. Glenzocimab for reperfusion in the setting of endovascular therapy for brain infarction: GREEN study. J Neurointerv Surg. 2025 Aug 27:jnis-2025-023606. doi: 10.1136/jnis-2025-023606. Online ahead of print. PMID 40866207